CLINICAL TRIAL: NCT04070326
Title: SPRING STUDY: An Open-Label, Multicenter, Phase 3 Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Lanadelumab for Prevention Against Acute Attacks of Hereditary Angioedema (HAE) in Pediatric Subjects 2 to <12 Years of Age
Brief Title: A Study of Lanadelumab to Prevent Hereditary Angioedema (HAE) Attacks in Children
Acronym: SPRING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHP643-301; 2018-002093-42 (EudraCT Number)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: Hereditary Angioedema
Keywords: Lanadelumab
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lanadelumab 150 mg: Age 2 to <6 Years (Experimental): Participants aged 2 to <6 years received lanadelumab subcutaneous (SC) injection at a dose of 150 milligrams (mg) for every 4 weeks (q4wks) over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B).
  Interventions: Drug: Lanadelumab
- Lanadelumab 150 mg: Age 6 to <12 Years (Experimental): Participants aged 6 to <12 years received lanadelumab SC injection at a dose of 150 mg for every 2 weeks (q2wks) over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B). Participants could switch to a dosing regimen of 150 mg q4wks in Treatment Period B at the investigator's discretion and sponsor's medical monitor approval, if they were well controlled (e.g., attack free) for 26 weeks with lanadelumab treatment in this study.Participants aged 6 to <12 years received lanadelumab SC injection at a dose of 150 mg for every 2 weeks (q2wks) over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B). Participants could switch to a dosing regimen of 150 mg q4wks in Treatment Period B at the investigator's discretion and sponsor's medical monitor approval, if they were well controlled (e.g., attack free) for 26 weeks with lanadelumab treatment in this study.
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — Participants will receive 150 mg dose of lanadelumab every 2 or 4 weeks, depending on the participants age, over the 52-week treatment period.
  Other Names: TAK-743; DX-2930; SHP643

SUMMARY:
The main aims of this study are to learn how lanadelumab moves through a child's body and if the children have any medical problems from lanadelumab. Other aims are to learn if prophylactic treatment with lanadelumab reduces the number and severity of HAE attacks in children, how lanadelumab affects the child's body, and if the children develop antibodies to lanadelumab.

The study doctors will treat acute HAE attacks according to their standard practice.

Participants will receive lanadelumab for up to 52 weeks. When they start treatment, participants will visit their clinic every week for the first 4 weeks. Then, they will visit their clinic every 4 weeks during treatment.

DETAILED DESCRIPTION:
This study will consists of 52-week treatment period and a 2 or 4-weeks follow-up period (depending on the treatment schedule). 52-week treatment period comprises of a 26-week treatment period A (Day 0 to Day 182) and a 26-week treatment period B (Day 183 to Day 364). Participants who complete treatment period A will immediately continue into treatment period B.

ELIGIBILITY:
Inclusion Criteria:

* Be a child (male or female) 2 to lesser than (<) 12 years of age at the time of screening.
* Documented diagnosis of HAE (Type I or II) based upon both of the following:

  1. Documented clinical history consistent with HAE (SC or mucosal, nonpruritic swelling episodes without accompanying urticarial).
  2. Diagnostic testing results obtained during screening from a sponsor- approved central laboratory that confirm C1-INH functional level < 40 percent (%) of the normal level. Participants with functional C1 esterase inhibitor (C1-INH) level 40-50% of the normal level may be enrolled if they also have a complement4 (C4) level below the normal range. With prior sponsor approval, participants may be retested during the baseline observation period if results are incongruent with clinical history or believed by the investigator to be confounded by recent complement1 (C1) inhibitor use.
* A historical baseline HAE attack rate of at least 1 attack per 3 months. Note: In addition, participants who experience greater than or equal to (>=)1.0 angioedema attacks per three months during the 12-week baseline observation period and who remain eligible per the inclusion criteria will enter the lanadelumab treatment period.
* Agree to adhere to the protocol-defined schedule of treatments, assessments, and procedures.
* Have a parent(s)/legal guardian who is informed of the nature of the study and can provide written informed consent for the child to participate in the study before any study-specific procedures are performed (with assent from the child when appropriate).
* Females of childbearing potential must agree to be abstinent or agree to comply with the applicable contraceptive requirements of this protocol through the duration of the study from screening through 70 days after the final study visit.

Exclusion Criteria:

* Concomitant diagnosis of another form of chronic, recurrent angioedema, such as acquired angioedema (AAE), HAE with normal C1-INH, idiopathic angioedema, or recurrent angioedema associated with urticaria.
* Dosing with an investigational drug or exposure to an investigational device within 4 weeks prior to screening.
* Be pregnant or breastfeeding.
* Have initiated androgen treatment (eg, stanozolol, danazol, oxandrolone, methyltestosterone, and testosterone) within 2 weeks prior to entering the observation period.
* Exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) within 4 weeks prior to screening.
* Have any active infectious illness or fever defined as an oral temperature greater than (>) 38 degree celsius (°C) (100.4 fahrenheit [°F]), tympanic > 38.5°C (101.3°F) , axillary > 38°C (100.4°F), or rectal/core > 38.5°C (101.3°F) within 24 hours prior to the first dose of study drug in treatment period A.
* Have any HAE attack that is not resolved prior to the first dose of study drug in treatment period A.
* Have any of the following liver function test abnormalities: alanine aminotransferase (ALT) > 3*upper limit of normal (ULN), or aspartate aminotransferase (AST) > 3*ULN, or total bilirubin > 2*ULN (unless the bilirubin elevation is a result of Gilbert's syndrome).
* Have any condition (any surgical or medical condition) that, in the opinion of the investigator or sponsor, may compromise their safety or compliance, preclude the successful conduct of the study, or interfere with interpretation of the results (eg, significant pre-existing illness or other major comorbidity that the investigator considers may confound the interpretation of study results).
* Participant has a known hypersensitivity to the investigational product or its components.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- United States (11):
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Institute Asthma and Allergy, Chevy Chase, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Hudson-Essex Allergy, Belleville, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Clinical Research Center of Charlotte, Charlotte, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Toledo Institute of Clinical Research Asthma & Allergy Center, Toledo, Ohio
  - AARA Research Center, Dallas, Texas
- Yang Medicine, Ottawa, Ontario, Canada
- Germany (3):
  - Charité - Universitätsmedizin Berlin., Berlin
  - Klinikum der Johann-Wolfgang Goethe-Universitat., Frankfurt
  - Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Semmelweis Egyetem., Budapest, Hungary
- Hospital Universitario La Paz. Paseo de la Castellana, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Maurer M, Lumry WR, Li HH, Aygoren-Pursun E, Busse PJ, Jacobs J, Nurse C, Ahmed MA, Watt M, Yu M; SPRING Investigators. Lanadelumab in Patients 2 to Less Than 12 Years Old With Hereditary Angioedema: Results From the Phase 3 SPRING Study. J Allergy Clin Immunol Pract. 2024 Jan;12(1):201-211.e6. doi: 10.1016/j.jaip.2023.09.009. Epub 2023 Sep 18. PMID 37730089
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab472e6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 24 participants were screened and 21 participants were enrolled in the study at 15 investigative sites in the United States, Canada, Spain, Hungary, and Germany from 19 August 2019 to 30 October 2021.
Pre-assignment Details: Enrolled participants were observed in 12-week Baseline Observation Period. Participants who experienced ≥1.0 angioedema attacks per 3 months during 12-week Baseline Observation Period and who remained eligible per inclusion criteria entered lanadelumab treatment period(TP). Pediatric participants aged 2 to <12 years received lanadelumab subcutaneous (SC) injection at a dose of 150 milligrams (mg) for every 4 weeks (q4wks) or for every 2 weeks (q2wks) based on age over 52-week Treatment Period.
Groups:
- Lanadelumab 150 mg: Age 2 to <6 Years: Participants aged 2 to <6 years received lanadelumab SC injection at a dose of 150 mg for q4wks over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B).
- Lanadelumab 150 mg: Age 6 to <12 Years: Participants aged 6 to <12 years received lanadelumab SC injection at a dose of 150 mg for q2wks over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B). Participants could switch to a dosing regimen of 150 mg q4wks in Treatment Period B at the investigator's discretion and sponsor's medical monitor approval, if they were well controlled (e.g., attack free) for 26 weeks with lanadelumab treatment in this study.
Period: Baseline Observation-12 Weeks Before TP
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Started | 4 | 17
Completed | 4 | 17
Not Completed | 0 | 0
Period: Treatment Period A (Weeks 1 to 26)
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Started | 4 | 17
Completed | 3 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 0
Period: Treatment Period B (Weeks 27 to 52)
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Started | 3 | 17
Completed | 3 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set consisted of all participants who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years | Total
Number analyzed (Participants) | 4 | 17 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.45 (0.843) | 8.68 (1.391) | 7.88 (2.134)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 2 | 7 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 15 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 16 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Including Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this investigational product or medicinal product. A SAE is any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose which results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, is an important medical event. Adverse events of special interest for this study are hypersensitivity reactions and disordered coagulation (hypercoagulability events and bleeding events).
Time Frame: Up to approximately 115 weeks
Population: The Safety Analysis Set consisted of all participants who received study drug. Overall number analyzed are participants presented by the actual treatment regimen. Because of dose modifications, some participants were treated with both dosing regimens and were counted in both treatment groups.
Measure: Count of Participants; unit: Participants
Groups:
- Lanadelumab 150 mg, q4wks: Participants received lanadelumab SC injection at a dose of 150 mg for q4wks with over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B).
- Lanadelumab 150 mg, q2wks: Participants received lanadelumab SC injection at a dose of 150 mg for q2wks over 52-week Treatment Period (26-week Treatment Period A and 26-week Treatment Period B).
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
Participants
  SAEs | 0 | 0
  AESIs | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities
Description: Laboratory values (chemistry, hematology, and coagulation) were to be considered clinically significant based on investigator's discretion.
Time Frame: Up to approximately 115 weeks
Population: The Safety Analysis Set consisted of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Measurements
Description: Vital signs included blood pressure, heart rate, body temperature, and respiratory rate.
Time Frame: Up to approximately 115 weeks
Population: The Safety Analysis Set consisted of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
Participants | 0 | 0

4. Primary Outcome: Plasma Concentrations of Lanadelumab Over The Treatment Period
Description: The plasma concentration of lanadelumab over treatment period was assessed.
Time Frame: Day 0 (Pre-dose), Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: The Pharmacokinetic (PK) Set included all participants in the Safety Analysis Set who have at least 1 evaluable post dose PK concentration value. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
nanograms per milliliter (ng/mL)
  Visit 1 Day 0 | 0.000 (0.0000) | 11.735 (39.2984)
  Visit 2 Day 4: number analyzed (Participants) | 3 | 14
  Visit 2 Day 4 | 32407.215 (9785.4332) | 20349.609 (12587.7085)
  Visit 3 Day 14 | 20443.818 (7800.4019) | 14589.883 (4734.4461)
  Visit 4 Day 28: number analyzed (Participants) | 4 | 14
  Visit 4 Day 28 | 10636.682 (6168.5347) | 21198.858 (8378.3961)
  Visit 8 Day 56: number analyzed (Participants) | 3 | 14
  Visit 8 Day 56 | 10433.382 (3345.1718) | 27751.659 (10048.7527)
  Visit 12 Day 84: number analyzed (Participants) | 3 | 14
  Visit 12 Day 84 | 14758.407 (8392.8620) | 24895.121 (11852.7671)
  Visit 16 Day 112: number analyzed (Participants) | 3 | 10
  Visit 16 Day 112 | 15020.780 (5730.4397) | 31053.260 (14012.6464)
  Visit 20 Day 140: number analyzed (Participants) | 3 | 12
  Visit 20 Day 140 | 13318.715 (4432.0728) | 26534.885 (11234.6051)
  Visit 24 Day 168: number analyzed (Participants) | 3 | 12
  Visit 24 Day 168 | 12189.214 (11367.4241) | 26166.340 (11070.0337)
  Visit 26 Day 182: number analyzed (Participants) | 3 | 11
  Visit 26 Day 182 | 25630.909 (11054.3701) | 25372.349 (8242.4858)
  Visit 28 Day 196: number analyzed (Participants) | 3 | 14
  Visit 28 Day 196 | 14293.013 (6014.0384) | 25238.600 (9921.4264)
  Visit 36 Day 252: number analyzed (Participants) | 3 | 16
  Visit 36 Day 252 | 23110.526 (18241.5743) | 19058.886 (12079.1976)
  Visit 44 Day 308: number analyzed (Participants) | 3 | 16
  Visit 44 Day 308 | 22687.442 (20911.9442) | 15774.463 (12043.0984)
  Visit 52 Day 364: number analyzed (Participants) | 3 | 15
  Visit 52 Day 364 | 27178.967 (24111.9243) | 17239.653 (11975.4861)
  Visit 56 Day 392 (End of Study Visit): number analyzed (Participants) | 2 | 14
  Visit 56 Day 392 (End of Study Visit) | 32400.148 (24303.4128) | 15689.458 (11811.7412)

5. Primary Outcome: Maximum Observed Concentration at Steady State (Cmax,ss) of Lanadelumab in Plasma
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: The PK Set included all participants in the Safety Analysis Set who have at least 1 evaluable post dose PK concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per mL (μg/mL)
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
micrograms per mL (μg/mL) | 37.7 (30.1) | 39.0 (39.2)

6. Primary Outcome: Average Concentration Over Dosing Interval at Steady State (Cavg,ss) of Lanadelumab in Plasma
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
μg/mL | 24.6 (34.0) | 33.2 (37.7)

7. Primary Outcome: Minimum Concentration at Steady State (Cmin,ss) of Lanadelumab in Plasma
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
µg/mL | 11.1 (46.5) | 24.8 (37.3)

8. Primary Outcome: Time to Reach Maximum Observed Concentration (Cmax) [Tmax] of Lanadelumab in Plasma
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
hours (h) | 122 [108 to 135] | 86.0 [66.0 to 137]

9. Primary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval at Steady State (AUCtau,ss) of Lanadelumab in Plasma
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg.day/mL
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
μg.day/mL | 690 (34.0) | 464 (37.7)

10. Primary Outcome: Terminal Half-life (t1/2) of Lanadelumab in Plasma
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
days | 11.7 [10.2 to 13.9] | 12.6 [9.59 to 27.3]

11. Primary Outcome: Apparent Clearance (CL/F) of Lanadelumab
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
L/h | 0.00906 (34.0) | 0.0135 (37.8)

12. Primary Outcome: Apparent Volume of Distribution (V/F) of Lanadelumab
Time Frame: Day 0 (Pre-dose), at any time pre-dose on Day 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
L | 3.63 (25.9) | 5.59 (39.2)

13. Secondary Outcome: Normalized Number of Investigator-Confirmed Hereditary Angioedema (HAE) Attacks During Overall Treatment Period
Description: Normalized number of investigator-confirmed HAE attacks during overall period are expressed as a monthly HAE attack rate. Investigator-confirmed HAE attack rate was calculated for each participant as number of investigator-confirmed HAE attacks occurring during given study period divided by the number of days the participant contributed to the period multiplied by 28 days. A HAE attack is defined as the symptoms or signs consistent with an attack in >=1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Day 0 (after start of study drug administration) through Day 364 (Week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
HAE attacks per month | 0.07 (0.219) | 0.08 (0.157)

14. Secondary Outcome: Normalized Number of Investigator-Confirmed HAE Attacks For Each Efficacy Evaluation Period Other Than the Overall Treatment Period
Description: Normalized number of investigator-confirmed HAE attacks during each efficacy evaluation period other than overall treatment period are expressed as a monthly HAE attack rate. Investigator-confirmed HAE attack rate was calculated for each participant as number of investigator-confirmed HAE attacks occurring during given study period divided by number of days participant contributed to period multiplied by 28 days. A HAE attack is defined as symptoms or signs consistent with an attack in at least 1 of following locations: peripheral angioedema (cutaneous swelling involving an extremity, face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
HAE attacks per month
  Overall Presumed Steady-state Period: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period | 0.09 (0.288) | 0.07 (0.143)
  Treatment Period A: number analyzed (Participants) | 4 | 17
  Treatment Period A | 0.15 (0.308) | 0.08 (0.207)
  Presumed Steady-state Period for Treatment Period A: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A | 0.25 (0.433) | 0.06 (0.192)
  Treatment Period B: number analyzed (Participants) | 10 | 18
  Treatment Period B | 0.28 (0.878) | 0.08 (0.142)

15. Secondary Outcome: Time to the First Investigator-Confirmed HAE Attack for Each Evaluation Period
Description: Time to first investigator-confirmed HAE attack (days) for each efficacy evaluation period was calculated from date and time of first dose of lanadelumab for that efficacy evaluation period to date and time of first investigator-confirmed HAE attack after first open-label dose for that efficacy evaluation period. A HAE attack is defined as symptoms or signs consistent with an attack in >=1 of following locations: peripheral angioedema (cutaneous swelling involving an extremity, face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of tongue, palate, uvula, or larynx). Kaplan-Meier Method was used for analysis.
Time Frame: Day 0 through Day 364, Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
days
  Treatment Period A | NA [NA to NA] — The median and 95% confidence interval (CI) were not evaluable due to low number of events. | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events.
  Presumed Steady-state Period for Treatment Period A: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events. | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events.
  Treatment Period B: number analyzed (Participants) | 10 | 18
  Treatment Period B | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events. | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events.
  Overall Treatment Period | NA [NA to NA] — The median and 95% CI were not avaluable due to low number of events. | NA [NA to NA] — The median and 95% CI were not avaluable due to low number of events.
  Overall Presumed Steady-state Period: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events. | NA [NA to NA] — The median and 95% CI were not evaluable due to low number of events.

16. Secondary Outcome: Normalized Number of HAE Attacks Requiring Acute Treatment for Each Efficacy Evaluation Period
Description: The normalized number of investigator-confirmed HAE attacks requiring acute treatment during each efficacy evaluation period are expressed as a monthly HAE attack rate. The investigator-confirmed HAE attack rate was calculated for each participant as the number of investigator-confirmed HAE attacks occurring during the given study period divided by the number of days the participant contributed to the period multiplied by 28 days. A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Day 0 through Day 364, Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
HAE attacks per month
  Overall Treatment Period | 0.07 (0.219) | 0.07 (0.140)
  Overall Presumed Steady-state Period: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period | 0.09 (0.288) | 0.06 (0.126)
  Treatment Period A: number analyzed (Participants) | 4 | 17
  Treatment Period A | 0.15 (0.308) | 0.07 (0.175)
  Presumed Steady-state Period for Treatment Period A: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A | 0.25 (0.433) | 0.04 (0.135)
  Treatment Period B: number analyzed (Participants) | 10 | 18
  Treatment Period B | 0.28 (0.878) | 0.06 (0.132)

17. Secondary Outcome: Normalized Number of Moderate or Severe Investigator-Confirmed HAE Attacks for Each Efficacy Evaluation Period
Description: The normalized number of moderate or severe investigator-confirmed HAE attacks requiring acute treatment during each efficacy evaluation period are expressed as a monthly HAE attack rate. The investigator-confirmed HAE attack rate was calculated for each participant as the number of investigator-confirmed HAE attacks occurring during the given study period divided by the number of days the participant contributed to the period multiplied by 28 days. A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Day 0 through Day 364, Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
HAE attacks per month
  Overall Treatment Period | 0.07 (0.219) | 0.07 (0.144)
  Overall Presumed Steady-state Period: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period | 0.09 (0.288) | 0.06 (0.125)
  Treatment Period A: number analyzed (Participants) | 4 | 17
  Treatment Period A | 0.15 (0.308) | 0.07 (0.175)
  Steady-state Period for Treatment Period A: number analyzed (Participants) | 3 | 17
  Steady-state Period for Treatment Period A | 0.25 (0.433) | 0.04 (0.135)
  Treatment Period B: number analyzed (Participants) | 10 | 18
  Treatment Period B | 0.3 (0.88) | 0.1 (0.13)

18. Secondary Outcome: Normalized Number of High Morbidity Investigator-Confirmed HAE Attacks for Each Efficacy Evaluation Period
Description: The normalized number of high morbidity investigator-confirmed HAE attacks requiring acute treatment during each efficacy evaluation period are expressed as a monthly HAE attack rate. The investigator-confirmed HAE attack rate was calculated for each participant as the number of investigator-confirmed HAE attacks occurring during the given study period divided by the number of days the participant contributed to the period multiplied by 28 days. A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Day 0 through Day 364, Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
HAE attacks per month
  Overall Treatment Period | 0.01 (0.044) | 0.01 (0.039)
  Overall Presumed Steady-state Period: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period | 0.02 (0.072) | 0.01 (0.039)
  Treatment Period A: number analyzed (Participants) | 4 | 17
  Treatment Period A | 0.04 (0.077) | 0.00 (0.000)
  Presumed Steady-state Period for Treatment Period A: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A | 0.08 (0.144) | 0.00 (0.000)
  Treatment Period B: number analyzed (Participants) | 10 | 18
  Treatment Period B | 0.00 (0.000) | 0.01 (0.039)

19. Secondary Outcome: Number of Participants With Characteristics of Investigator-Confirmed HAE Attacks for Each Efficacy Evaluation Period
Description: Characteristics of investigator-confirmed HAE attacks for each efficacy evaluation period included duration, severity, attack location, and rescue medication use. A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). Only categories with data are reported.
Time Frame: Day 0 through Day 364, Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
Participants
  Treatment Period A: Mean HAE attack duration: 0 hour: number analyzed (Participants) | 4 | 17
  Treatment Period A: Mean HAE attack duration: 0 hour | 3 | 14
  Treatment Period A: Mean HAE attack duration: <12 hours | 1 | 2
  Treatment Period A: Mean HAE attack duration: >24-48 hours: number analyzed (Participants) | 4 | 17
  Treatment Period A: Mean HAE attack duration: >24-48 hours | 0 | 1
  Treatment Period A: Maximum HAE attack severity: No attack: number analyzed (Participants) | 4 | 17
  Treatment Period A: Maximum HAE attack severity: No attack | 3 | 14
  Treatment Period A: Maximum HAE attack severity: Moderate: number analyzed (Participants) | 4 | 17
  Treatment Period A: Maximum HAE attack severity: Moderate | 0 | 3
  Treatment Period A: Maximum HAE attack severity: Severe: number analyzed (Participants) | 4 | 17
  Treatment Period A: Maximum HAE attack severity: Severe | 1 | 0
  Presumed Steady-state Period for Treatment Period A: Mean HAE attack duration: 0 hour: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Mean HAE attack duration: 0 hour | 2 | 15
  Presumed Steady-state Period for Treatment Period A: Mean HAE attack duration: <12 hours: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Mean HAE attack duration: <12 hours | 1 | 1
  Presumed Steady-state Period for Treatment Period A: Mean HAE attack duration: >24-48 hours: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Mean HAE attack duration: >24-48 hours | 0 | 1
  Presumed Steady-state Period for Treatment Period A: Maximum HAE attack severity: No attack: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Maximum HAE attack severity: No attack | 2 | 15
  Presumed Steady-state Period for Treatment Period A: Maximum HAE attack severity: Moderate: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Maximum HAE attack severity: Moderate | 0 | 2
  Presumed Steady-state Period for Treatment Period A: Maximum HAE attack severity: Severe: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Maximum HAE attack severity: Severe | 1 | 0
  Treatment Period B: Mean HAE attack duration: 0 hour: number analyzed (Participants) | 10 | 18
  Treatment Period B: Mean HAE attack duration: 0 hour | 9 | 13
  Treatment Period B: Mean HAE attack duration: >0-<12 hours: number analyzed (Participants) | 10 | 18
  Treatment Period B: Mean HAE attack duration: >0-<12 hours | 1 | 3
  Treatment Period B: Mean HAE attack duration: 12-24 hours: number analyzed (Participants) | 10 | 18
  Treatment Period B: Mean HAE attack duration: 12-24 hours | 0 | 1
  Treatment Period B: Mean HAE attack duration: >48 hours: number analyzed (Participants) | 10 | 18
  Treatment Period B: Mean HAE attack duration: >48 hours | 0 | 1
  Treatment Period B: Maximum HAE attack severity: No attack: number analyzed (Participants) | 10 | 18
  Treatment Period B: Maximum HAE attack severity: No attack | 9 | 13
  Treatment Period B: Maximum HAE attack severity: Moderate: number analyzed (Participants) | 10 | 18
  Treatment Period B: Maximum HAE attack severity: Moderate | 1 | 4
  Treatment Period B: Maximum HAE attack severity: Severe: number analyzed (Participants) | 10 | 18
  Treatment Period B: Maximum HAE attack severity: Severe | 0 | 1
  Overall Treatment Period: Mean HAE attack duration: 0 hour | 10 | 13
  Overall Treatment Period: Mean HAE attack duration: >0-<12 hours | 1 | 4
  Overall Treatment Period: Mean HAE attack duration: >24-48 hours | 0 | 1
  Overall Treatment Period: Maximum HAE attack severity: No attack | 10 | 13
  Overall Treatment Period: Maximum HAE attack severity: Moderate | 0 | 4
  Overall Treatment Period: Maximum HAE attack severity: Severe | 1 | 1
  Overall Presumed Steady-state Period: Mean HAE attack duration: 0 hour: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Mean HAE attack duration: 0 hour | 9 | 13
  Overall Presumed Steady-state Period: Mean HAE attack duration: >0-<12 hours: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Mean HAE attack duration: >0-<12 hours | 1 | 4
  Overall Presumed Steady-state Period: Mean HAE attack duration: >48 hours: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Mean HAE attack duration: >48 hours | 0 | 1
  Overall Presumed Steady-state Period: Maximum HAE attack severity: No attack: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Maximum HAE attack severity: No attack | 9 | 13
  Overall Presumed Steady-state Period: Maximum HAE attack severity: Moderate: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Maximum HAE attack severity: Moderate | 0 | 4
  Overall Presumed Steady-state Period: Maximum HAE attack severity: Severe: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Maximum HAE attack severity: Severe | 1 | 1
  Treatment Period A: HAE Primary Attack Location: Peripheral: number analyzed (Participants) | 4 | 17
  Treatment Period A: HAE Primary Attack Location: Peripheral | 1 | 2
  Treatment Period A: HAE Primary Attack Location: Abdominal: number analyzed (Participants) | 4 | 17
  Treatment Period A: HAE Primary Attack Location: Abdominal | 1 | 1
  Treatment Period A: HAE Attack Derived Location: Peripheral: number analyzed (Participants) | 4 | 17
  Treatment Period A: HAE Attack Derived Location: Peripheral | 1 | 2
  Treatment Period A: HAE Attack Derived Location: Abdominal: number analyzed (Participants) | 4 | 17
  Treatment Period A: HAE Attack Derived Location: Abdominal | 1 | 1
  Treatment Period A: Rescue Medication Use: No Use: number analyzed (Participants) | 4 | 17
  Treatment Period A: Rescue Medication Use: No Use | 0 | 1
  Treatment Period A: Rescue Medication Use: Icatibant: number analyzed (Participants) | 4 | 17
  Treatment Period A: Rescue Medication Use: Icatibant | 0 | 1
  Treatment Period A: Rescue Medication Use: C1-INH (Nano-filtered C1-INH): number analyzed (Participants) | 4 | 17
  Treatment Period A: Rescue Medication Use: C1-INH (Nano-filtered C1-INH) | 0 | 1
  Treatment Period A: Rescue Medication Use: C1-INH (Plasma-derived): number analyzed (Participants) | 4 | 17
  Treatment Period A: Rescue Medication Use: C1-INH (Plasma-derived) | 1 | 1
  Presumed Steady-state Period for Treatment Period A: HAE Primary Attack Location: Peripheral: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: HAE Primary Attack Location: Peripheral | 0 | 2
  Presumed Steady-state Period for Treatment Period A: HAE Primary Attack Location: Abdominal: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: HAE Primary Attack Location: Abdominal | 1 | 0
  Presumed Steady-state Period for Treatment Period A: HAE Attack Derived Location: Peripheral: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: HAE Attack Derived Location: Peripheral | 0 | 2
  Presumed Steady-state Period for Treatment Period A: HAE Attack Derived Location: Abdominal: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: HAE Attack Derived Location: Abdominal | 1 | 0
  Presumed Steady-state Period for Treatment Period A: Rescue Medication Use: No Use: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Rescue Medication Use: No Use | 0 | 1
  Presumed Steady-state Period for Treatment Period A: Rescue Medication Use: Icatibant: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A: Rescue Medication Use: Icatibant | 0 | 1
  Presumed Steady-state Period for Treatment Period A:Rescue Medication Use:Plasma-derived C1-INH: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A:Rescue Medication Use:Plasma-derived C1-INH | 1 | 1
  Treatment Period B: HAE Primary Attack Location: Peripheral: number analyzed (Participants) | 10 | 18
  Treatment Period B: HAE Primary Attack Location: Peripheral | 0 | 3
  Treatment Period B: HAE Primary Attack Location: Abdominal: number analyzed (Participants) | 10 | 18
  Treatment Period B: HAE Primary Attack Location: Abdominal | 1 | 4
  Treatment Period B: HAE Attack Derived Location: Peripheral: number analyzed (Participants) | 10 | 18
  Treatment Period B: HAE Attack Derived Location: Peripheral | 0 | 3
  Treatment Period B: HAE Attack Derived Location: Abdominal: number analyzed (Participants) | 10 | 18
  Treatment Period B: HAE Attack Derived Location: Abdominal | 1 | 4
  Treatment Period B: Rescue Medication Use: No Use: number analyzed (Participants) | 10 | 18
  Treatment Period B: Rescue Medication Use: No Use | 0 | 2
  Treatment Period B: Rescue Medication Use: Icatibant: number analyzed (Participants) | 10 | 18
  Treatment Period B: Rescue Medication Use: Icatibant | 0 | 2
  Treatment Period B: Rescue Medication Use: C1-INH (Plasma-derived C1-INH): number analyzed (Participants) | 10 | 18
  Treatment Period B: Rescue Medication Use: C1-INH (Plasma-derived C1-INH) | 1 | 2
  Overall Treatment Period: HAE Primary Attack Location: Peripheral | 1 | 3
  Overall Treatment Period: HAE Primary Attack Location: Abdominal | 1 | 4
  Overall Treatment Period: HAE Attack Derived Location: Peripheral | 1 | 3
  Overall Treatment Period: HAE Attack Derived Location: Abdominal | 1 | 4
  Overall Treatment Period: Rescue Medication Use: No Use | 0 | 3
  Overall Treatment Period: Rescue Medication Use: Icatibant | 0 | 2
  Overall Treatment Period: Rescue Medication Use: C1-INH (Nano-filtered C1-INH) | 0 | 1
  Overall Treatment Period: Rescue Medication Use: C1-INH (Plasma-derived C1-INH) | 1 | 2
  Overall Presumed Steady-state Period: HAE Primary Attack Location: Peripheral: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: HAE Primary Attack Location: Peripheral | 0 | 3
  Overall Presumed Steady-state Period: HAE Primary Attack Location: Abdominal: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: HAE Primary Attack Location: Abdominal | 1 | 4
  Overall Presumed Steady-state Period: HAE Attack Derived Location: Peripheral: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: HAE Attack Derived Location: Peripheral | 0 | 3
  Overall Presumed Steady-state Period: HAE Attack Derived Location: Abdominal: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: HAE Attack Derived Location: Abdominal | 1 | 4
  Overall Presumed Steady-state Period: Rescue Medication Use: No Use: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Rescue Medication Use: No Use | 0 | 3
  Overall Presumed Steady-state Period: Rescue Medication Use: Icatibant: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Rescue Medication Use: Icatibant | 0 | 2
  Overall Presumed Steady-state Period: Rescue Medication Use: C1-INH (Plasma-derived C1-INH): number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period: Rescue Medication Use: C1-INH (Plasma-derived C1-INH) | 1 | 2

20. Secondary Outcome: Number of Participants With HAE Attack-Free Status for Each Evaluation Period
Description: A HAE attack is defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Day 0 through Day 364, Day 0 through Day 182, Day 70 through Day 182, Day 183 through Day 364, Day 70 through Day 364
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
Number analyzed (Participants) | 11 | 18
Participants
  Treatment Period A: number analyzed (Participants) | 4 | 17
  Treatment Period A | 3 | 14
  Presumed Steady-state Period for Treatment Period A: number analyzed (Participants) | 3 | 17
  Presumed Steady-state Period for Treatment Period A | 2 | 15
  Treatment Period B: number analyzed (Participants) | 10 | 18
  Treatment Period B | 9 | 13
  Overall Treatment Period | 10 | 13
  Overall Presumed Steady-state Period: number analyzed (Participants) | 10 | 18
  Overall Presumed Steady-state Period | 9 | 13

21. Secondary Outcome: Plasma Kallikrein (pKal) Activity
Description: pKal activity was measured by biomarker cleaved high molecular weight kininogen (cHMWK) level to assess pharmacodynamics of lanadelumab.
Time Frame: Day 0 (Pre-dose), at any time on Days 4, 14, 28, 56, 84, 112, 140, 168, 182 196, 252, 308, 364 and 392
Population: The Pharmacodynamic (PD) Set included all participants in the Safety Analysis Set who have at least 1 evaluable post dose PD value. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: percentage of cHMWK
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
percentage of cHMWK
  Visit 1 Day 0: number analyzed (Participants) | 4 | 16
  Visit 1 Day 0 | 30.2500 (13.61017) | 45.6438 (25.79470)
  Visit 2 Day 4: number analyzed (Participants) | 3 | 14
  Visit 2 Day 4 | 16.4000 (8.94036) | 32.2857 (17.89606)
  Visit 3 Day 14 | 9.5750 (4.05740) | 25.7176 (11.75565)
  Visit 4 Day 28: number analyzed (Participants) | 4 | 14
  Visit 4 Day 28 | 18.8500 (14.15968) | 26.1571 (11.76616)
  Visit 8 Day 56: number analyzed (Participants) | 3 | 15
  Visit 8 Day 56 | 15.1333 (12.95582) | 24.6267 (14.28963)
  Visit 12 Day 84: number analyzed (Participants) | 3 | 14
  Visit 12 Day 84 | 18.2333 (17.91768) | 24.7214 (12.84339)
  Visit 16 Day 112: number analyzed (Participants) | 3 | 12
  Visit 16 Day 112 | 10.7333 (5.48118) | 18.0000 (11.05992)
  Visit 20 Day 140: number analyzed (Participants) | 3 | 12
  Visit 20 Day 140 | 15.2000 (16.96202) | 16.3417 (12.53841)
  Visit 24 Day 168: number analyzed (Participants) | 3 | 12
  Visit 24 Day 168 | 21.9000 (20.71545) | 19.6167 (16.61762)
  Visit 26 Day 182: number analyzed (Participants) | 3 | 11
  Visit 26 Day 182 | 17.9000 (14.29021) | 18.6818 (10.54332)
  Visit 28 Day 196: number analyzed (Participants) | 3 | 14
  Visit 28 Day 196 | 9.2000 (2.52389) | 14.6571 (7.29939)
  Visit 36 Day 252: number analyzed (Participants) | 3 | 15
  Visit 36 Day 252 | 15.2000 (13.16397) | 16.3067 (10.26008)
  Visit 44 Day 308: number analyzed (Participants) | 3 | 16
  Visit 44 Day 308 | 13.5333 (7.24316) | 23.2750 (15.23577)
  Visit 52 Day 364: number analyzed (Participants) | 3 | 15
  Visit 52 Day 364 | 10.7333 (2.87112) | 14.4733 (8.51448)
  Visit 56 Day 392 EOS: number analyzed (Participants) | 3 | 14
  Visit 56 Day 392 EOS | 10.9000 (3.15753) | 19.4286 (14.57677)

22. Secondary Outcome: Number of Participants With Immunogenicity Status as Positive or Negative
Description: Immunogenicity was measured based on the presence or absence of neutralizing or non-neutralizing Anti-drug Antibody (ADA) in plasma.
Time Frame: Day 0 (Pre-dose), Days 28, 84, 140, 182, 196, 252, 308, 364 and 392
Population: The Safety Analysis Set consisted of all participants who received study drug. Number analyzed are the number of participants with data available for given category.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 150 mg: Age 2 to <6 Years | Lanadelumab 150 mg: Age 6 to <12 Years
Number analyzed (Participants) | 4 | 17
Participants
  Baseline (Day 0): ADA Negative | 4 | 17
  Baseline (Day 0): ADA Positive | 0 | 0
  Baseline (Day 0): ADA Positive (Neutralizing) | 0 | 0
  Baseline (Day 0): ADA Positive (Non-neutralizing) | 0 | 0
  Visit 4 Day 28: ADA Negative: number analyzed (Participants) | 4 | 14
  Visit 4 Day 28: ADA Negative | 4 | 13
  Visit 4 Day 28: ADA Positive: number analyzed (Participants) | 4 | 14
  Visit 4 Day 28: ADA Positive | 0 | 1
  Visit 4 Day 28: ADA Positive (Neutralizing): number analyzed (Participants) | 4 | 14
  Visit 4 Day 28: ADA Positive (Neutralizing) | 0 | 0
  Visit 4 Day 28: ADA Positive (Non-neutralizing): number analyzed (Participants) | 4 | 14
  Visit 4 Day 28: ADA Positive (Non-neutralizing) | 0 | 1
  Overall Treatment Period A: ADA Negative: number analyzed (Participants) | 4 | 16
  Overall Treatment Period A: ADA Negative | 4 | 13
  Overall Treatment Period A: ADA Positive: number analyzed (Participants) | 4 | 16
  Overall Treatment Period A: ADA Positive | 0 | 3
  Overall Treatment Period A: ADA Positive (Neutralizing) | 0 | 1
  Overall Treatment Period A: ADA Positive (Non-neutralizing) | 0 | 3
  Overall Treatment Period B: ADA Negative: number analyzed (Participants) | 3 | 16
  Overall Treatment Period B: ADA Negative | 3 | 15
  Overall Treatment Period B: ADA Positive: number analyzed (Participants) | 3 | 16
  Overall Treatment Period B: ADA Positive | 0 | 1
  Overall Treatment Period B: ADA Positive (Neutralizing): number analyzed (Participants) | 3 | 16
  Overall Treatment Period B: ADA Positive (Neutralizing) | 0 | 0
  Overall Treatment Period B: ADA Positive (Non-neutralizing): number analyzed (Participants) | 3 | 16
  Overall Treatment Period B: ADA Positive (Non-neutralizing) | 0 | 1
  Overall Study Period: ADA Negative: number analyzed (Participants) | 4 | 16
  Overall Study Period: ADA Negative | 4 | 13
  Overall Study Period: ADA Positive: number analyzed (Participants) | 4 | 16
  Overall Study Period: ADA Positive | 0 | 3
  Overall Study Period: ADA Positive (Neutralizing): number analyzed (Participants) | 4 | 16
  Overall Study Period: ADA Positive (Neutralizing) | 0 | 1
  Overall Study Period: ADA Positive (Non-neutralizing): number analyzed (Participants) | 4 | 16
  Overall Study Period: ADA Positive (Non-neutralizing) | 0 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 115 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Overall number at risk are participants presented by the actual treatment regimen. Because of dose modifications, some participants were treated with both dosing regimens and were counted in both treatment groups.
Arm/Group | Lanadelumab 150 mg, q4wks | Lanadelumab 150 mg, q2wks
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/18
Other Adverse Events (participants affected / at risk) | 6/11 | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanadelumab 150 mg, q4wks (N=11) | Lanadelumab 150 mg, q2wks (N=18)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (12) | 6 (76)
Injection site erythema (General disorders) | 2 (8) | 2 (21)
Injection site swelling (General disorders) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Administration site pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Injection site injury (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Adenoiditis (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (3) | 3 (13)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (2)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (4):
  • Study Protocol: Original Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT04070326/Prot_000.pdf
  • Study Protocol: Amendment 1 (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT04070326/Prot_001.pdf
  • Study Protocol: Amendment 2 (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT04070326/Prot_002.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT04070326/SAP_003.pdf